CLINICAL TRIAL: NCT04305470
Title: A Phase 3 Multicenter Study of Gleolan (Aminolevulinic Acid Hydrochloride) to Enhance Visualization of Tumor in Patients With Newly Diagnosed or Recurrent Meningiomas
Brief Title: Gleolan for Visualization of Newly Diagnosed or Recurrent Meningioma
Acronym: MEN-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NX Development Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NXDC-MEN-301
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Meningioma
Keywords: ALA; fluorescence guided surgery; Gleolan; meningioma
MeSH Terms: conditions — Meningioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Phase 3, open-label, single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Open-label, single-arm
  Interventions: Drug: Gleolan (Aminolevulinic Acid Hydrochloride/ALA/ALA-HCI)

INTERVENTIONS:
Drug: Gleolan (Aminolevulinic Acid Hydrochloride/ALA/ALA-HCI) — One time oral dose on day of surgery (20 mg/kg bodyweight)

SUMMARY:
This Phase 3 open-label single-arm study is designed to investigate the safety, diagnostic performance, and clinical usefulness of Gleolan for the real time detection and visualization of meningiomas during tumor resection surgery. The study is planned to run for 15 months with individual study participation lasting for approximately 2 months.

DETAILED DESCRIPTION:
This Phase 3 open-label single-arm study is designed to investigate the safety, diagnostic performance, and clinical usefulness of the imaging agent Gleolan™ (Aminolevulinic Acid Hydrochloride, ALA HCl, ALA, 5-ALA), an orally administered imaging agent for the real time detection and visualization of meningiomas during tumor resection surgery. ALA is a prodrug that is metabolized intracellularly to form the fluorescent molecule Protoporphyrin IX (PpIX). The exogenous application of ALA leads to a highly selective accumulation of PpIX in tumor cells. Following excitation with blue light (BL) (λ = 375 - 440 nm), the PpIX, which has accumulated selectively in tumor tissue, emits a red-violet light. This phenomenon allows for the real-time visualization of tumor tissue during resection surgery.

Patients about to undergo resection for suspected meningioma [World Health Organization (WHO) Grade I, II, III] will be screened and informed consent will be obtained prior to surgery and prior to study participation. Eligible study participants will receive an oral solution of Gleolan (20 mg/kg body weight) 3 hours, (target range 2-4 hours) prior to anesthesia, and then undergo surgery for meningioma resection. During the surgery, the surgeon will use a microscope equipped with WL and BL for visualization of Gleolan-induced PpIX fluorescence for the selection of protocol-driven tissue locations and to assess fluorescence status.

Study participants will be evaluated within 48 hours post procedure, 2 weeks post procedure, and 6 weeks post procedure for study safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. A pre-operative MRI within ≥ 90 days of study enrollment documenting a suspected meningioma or suspected recurrence of a meningioma for which a meningioma resection is indicated and has been planned.
2. Adult age ≥ 18 years.
3. Patient must have normal organ and bone marrow function and be appropriate surgical candidates per site SOC.
4. Patient must have recording of each parameter as defined below:

   Bilirubin Below upper limit of normal AST (SGOT) < 2.5 X institutional upper limit of normal ALT (SGPT) < 2.5 X institutional upper limit of normal Creatinine Below upper limit of normal OR Creatinine clearance >60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
5. The patient must demonstrate the ability to understand the informed consent document and the willingness and ability to sign a written informed consent document. The study consent documents will be prepared in English and German and Spanish. Translation for non-English, non-German, or non-Spanish speaking participants will be provided as appropriate by institution, as required.
6. WOCBP and men participating must agree to use highly effective forms of contraception, and men must also agree not to donate sperm for the duration of treatment, and for at least 42 days after the one time use of the study drug.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical/biologic composition to Gleolan.
2. Known or documented personal or family history of porphyria.
3. Uncontrolled concurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness.
4. Patient has had a meningioma resection or radiation treatment within 90 days of informed consent.
5. Social or medical situations that would limit compliance with study requirements (e.g. ability to travel for follow-up or inability to obtain appropriate pre-op MRI (e.g. cardiac pacemaker).
6. Women who are pregnant or plan to become pregnant during study participation.
7. Prior history of gastrointestinal perforation, diverticulitis, and or/peptic ulcer disease within 90 days of informed consent.
8. Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding treatment or within 5 plasma half-life of the preceding study drug, whatever is longer.
9. Simultaneous use of other potentially phototoxic substances (St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulphonamides, quinolones and tetracyclines), and topical preparations containing ALA for 24 hours during the perioperative period (see MOPS for detailed list).
10. Unwillingness by patient to sign consent or return for subsequent visits following surgery.
11. Any condition that in the opinion of the Investigator would exclude the patient as a viable candidate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who have at least one indeterminate tissue or unexpected fluorescent End of Surgery (EOS) tissue where Gleolan-induced PpIX fluorescence status is consistent with histology. | Surgery (Day 1)
  Per Protocol Population

SECONDARY OUTCOMES:
Positive Predicted Value (PPV) of Gleolan-induced PpIX fluorescence of the single bulk tumor tissue obtained from each study participant | Surgery (Day 1)
  Per Protocol Population
Diagnostic accuracy of Gleolan-induced PpIX fluorescence among indeterminate tissue and unexpected fluorescent EOS tissue locations is at least 20% greater than the diagnostic accuracy of the surgeons' assessment. | Surgery (Day 1)
  Biopsy Efficacy Analysis Population
Diagnostic performance of Gleolan-induced PpIX fluorescence will be computed for indeterminate tissue biopsies, unexpected fluorescent EOS tissue biopsies. | Surgery (Day 1)
  Biopsy Efficacy Analysis Population
The concordance between the Surgeon and Adjudication Panel assessment of white light (WL) visualization visualization to identify tissue as likely or unlikely to be meningioma among indeterminate tissues. | Surgery (Day 1)
  Biopsy Efficacy Analysis Population
The concordance between the Surgeon and Adjudication Panel assessment of blue light (BL) visualization to identify fluorescence status of indeterminate tissues. | Surgery (Day 1)
  Biopsy Efficacy Analysis Population

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, MD, Principal Investigator — Universitätsklinikum Münster; Bernard Bendok, MD, Principal Investigator — Mayo Clinic
Locations (17):
- United States (15):
  - Mayo Clinic, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Keck Hospital of USC, Los Angeles, California
  - Providence St. Joseph Hospital, Orange, California
  - Swedish Medical Center, Englewood, Colorado
  - University of Miami, Coral Gables, Florida
  - Baptist Health South Florida, Miami, Florida
  - Southern Illinois University, Springfield, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - NYU Langone Health, Brooklyn, New York
  - University of Pennsylvania- Penn Medicine, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - MD Anderson, Houston, Texas
- Medical University of Vienna, Vienna, Austria
- University Hospital Münster, Münster, Germany